CLINICAL TRIAL: NCT03846258
Title: High Versus Low Bicarbonate Bath in Critically-ill Patients Receiving Continuous Renal Replacement Therapy: a Pragmatic Randomized Control Trial
Brief Title: High Versus Low Bicarbonate Bath in Critically-ill Patients Receiving Continuous Renal Replacement Therapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to the fact that we were unable to find subjects who met all inclusion and exclusion criteria it was determined to withdraw this study.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kianoush B. Kashani, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-010147
Record Dates: First submitted 2019-02-14; First posted 2019-02-19 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Metabolic Acidosis; Acute Kidney Injury; Acute Kidney Failure
MeSH Terms: conditions — Acidosis; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low bicarbonate arm (22 mmol/L) (Active Comparator): PHOXILLUM solutions are used as a replacement solution in Continuous Renal Replacement Therapy. The one to be used in this study has bicarbonate concentration of 22 mmol/L.
  Interventions: Drug: Low bicarbonate solution (22 mmol/L)
- High Bicarbonate (32 mmol/L) (Active Comparator): PrismaSATE is another replacement solution used in Continuous Renal Replacement Therapy. The one to be used in this study has bicarbonate concentration of 32 mmol/L.
  Interventions: Drug: High Bicarbonate solution (32 mmol/L)

INTERVENTIONS:
Drug: Low bicarbonate solution (22 mmol/L) — Participants randomized to this arm will be started on CRRT using Phoxillum as the replacement fluid.
  Other Names: Phoxillum
  Arms: Low bicarbonate arm (22 mmol/L)
Drug: High Bicarbonate solution (32 mmol/L) — Participants randomized to this arm will be started on CRRT using Prismasate as the replacement fluid.
  Other Names: Prismasate
  Arms: High Bicarbonate (32 mmol/L)

SUMMARY:
Researchers are trying to determine which dialysis solution, low bicarbonate fluid (22 mmol/L) or high bicarbonate fluid (32 mmol/L), is better in subjects with acute kidney injury (acute kidney failure) and metabolic acidosis that are admitted to the intensive care unit and require continuous renal replacement therapy (also known as continuous dialysis).

DETAILED DESCRIPTION:
This is a prospective randomized trial that will be conducted at Mayo Clinic in Rochester Minnesota. It will be based on Good Clinical Practice Standards and performed under IRB supervision. This will be a pragmatic clinical trial due to the nature of the intervention and short interval for making a clinical decision. While dialysis in general is valid in cases of severe AKI and metabolic acidosis, there remains uncertainty as to which replacement fluid to use. In one retrospective study, using high bicarbonate replacement fluid was associated with worse outcomes, even after accounting for several important confounders. While this intervention is valid in cases of severe metabolic acidosis (pH<7), there has not been much data to support the use of either intervention in cases of any metabolic acidosis in general.

While both interventions are equally valid, to our knowledge, there is no randomized clinical trial evaluating the difference of either intervention on outcomes. There is limited evidence in the literature on benefit or harm associated with either of the interventions on the outcomes thus generating a clinical equipoise. This pivotal study should help guide nephrologists and intensivists on the appropriate prescription of CRRT.

ELIGIBILITY:
Inclusion Criteria

* Adult patients (≥ 18 years of age)
* Ability to obtain informed consent, either from patient or legally authorized representative (LAR)
* Diagnosis of AKI according to KDIGO definition [an increase in serum creatinine concentration of greater than or equal to 0.3 mg/dL within the first 48 hours of injury, a relative increase in serum creatinine of greater than or equal to 50% (1.5-fold from baseline) within the first 7 days of injury, or a reduction in urine output (<0.5 mL/kg/h for more than 6 hours)]
* CRRT initiated for the first time during current ICU admission.
* Bicarbonate ≤ 22 mEq/L
* Arterial pH between 7.05 and 7.25(if an ABG is not available, venous pH must be between 7.00 and 7.20)

Exclusion Criteria

* Pregnancy (women of child-bearing potential must have a negative pregnancy test)
* Diagnosis of End-Stage renal disease and receiving Hemodialysis or peritoneal dialysis prior to ICU admission (this information will be easily obtained by the nephrology team)
* Arterial pH <7.05 or >7.25 (if an ABG is not available, Venous pH <7.00 or >7.20)
* Potassium level >6.0 mmol/L
* Severe acute liver failure meeting all the following criteria):

  * INR >2
  * AST/ALT more than 500 U/L and
  * Bilirubin more than 12 mg/dL)
* Previous enrollment in this study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 120 days
  Discharge status: death

SECONDARY OUTCOMES:
Time to achieve pH >7.3 | 30 days
  The number of hours it took each participant to have an arterial pH of >7.3 or a venous pH > 7.35 following CRRT initiation
Major Adverse Kidney events | 120 Days
  Composite outcome of death, persistent kidney dysfunction (creatinine more than 1.5 times baseline) or need for renal replacement therapy at specified time intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Kianoush B Kashani, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No